CLINICAL TRIAL: NCT07012434
Title: Exploring the Mechanisms of Postoperative Delirium in Cirrhotic Patients Through Multi-Omics Integrative Analysis: An Observational Study
Brief Title: Exploring the Mechanisms of Postoperative Delirium in Cirrhotic Patients Through Multi-Omics Integrative Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Peng Li, Deputy Director, Anesthesia and Surgery Center, Sichuan Provincial People's Hospital
Other Study IDs: SPPH2025381
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis
Keywords: Postoperative delirium; gut microbiota dysbiosis; metabolomics
MeSH Terms: conditions — Liver Cirrhosis; Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and anal swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with liver cirrhosis scheduled for upper abdominal surgery
- Patients without liver cirrhosis scheduled for upper abdominal surgery

SUMMARY:
This study looks at memory problems after surgery in people with liver disease. We want to know how often these problems happen and what might cause them. The main question it aims to answer is:

1. Do people with liver disease have more memory problems after stomach surgery than people without liver disease? If yes, how much more often?
2. Are changes in stomach bacteria and body chemicals related to these memory problems?

Who can join:

* Adults getting stomach surgery
* Both people with and without liver disease

What participants will do:

* Take memory tests before and after surgery
* Give stool (poop) and blood samples before and after surgery

Why this matters:

Memory problems after surgery can make recovery harder. If we find that stomach bacteria or body chemicals are involved, doctors might find new ways to prevent these problems in people with liver disease.

DETAILED DESCRIPTION:
Liver cirrhosis is one of the most prevalent global diseases, ranking as the 11th leading cause of death worldwide with approximately 1 million annual fatalities. China has an estimated 300 million patients with liver diseases, including 7 million cirrhosis cases, accounting for 11% of global cirrhosis-related mortality. Previous studies report that approximately 1 in 10 cirrhosis patients require hepatic or non-hepatic surgical interventions during their final two years of life. With advancements in perioperative techniques including surgery, anesthesia, critical care, and nursing, non-hepatic surgeries for cirrhotic patients have become increasingly common.

The major postoperative complications in cirrhotic patients include coma, hepatic failure, sepsis, hemorrhage, thrombosis, and renal failure, among which coma represents the most frequent complication. These findings highlight the critical scientific importance of reducing postoperative complications in cirrhotic patients, particularly neurological complications.

Postoperative delirium (POD) refers to delirium occurring within one week after surgical procedures, with characteristic temporal features predominantly manifesting 24-72 hours postoperation. POD adversely impacts both short- and long-term patient outcomes. Studies demonstrate that POD patients face 2-3 times higher risk of other postoperative complications, 2-3 times increased perioperative mortality risk and prolonged hospitalization. Long-term follow-up studies reveal that POD patients exhibit increased incidence of postoperative cognitive dysfunction, reduced quality of life and higher long-term mortality rates. Cirrhotic patients frequently present with overt or subclinical cognitive impairment. Surgical intervention in this population may exacerbate neurological dysfunction, potentially explaining the significantly elevated risk of postoperative neurological complications. The commonly observed gut microbiota dysbiosis and metabolic disturbances in cirrhotic patients may play pivotal roles in this process.

This study aims to compare POD incidence and perioperative cognitive function changes between cirrhotic and non-cirrhotic patients undergoing upper abdominal surgery, and investigate the role of gut microbiota dysbiosis and metabolic abnormalities in POD pathogenesis among cirrhotic patients through integrated microbiome-metabolome analysis. The findings may provide valuable insights into the mechanisms and potential therapeutic approaches for cognitive dysfunction in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years
2. Patients with or without liver cirrhosis scheduled for upper abdominal surgery due to various clinical indications
3. Ability to comply with the study protocol and provide informed consent

Exclusion Criteria:

1. Comorbid severe cardiac, pulmonary, or renal diseases
2. Patients with mental status incompatible with study participation, including:

   * Psychiatric disorders
   * Inability to communicate clearly
3. Any condition preventing effective communication or cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients scheduled for surgical treatment at Sichuan Provincial People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium within 7 days after upper abdominal surgery in patients with liver cirrhosis. | within 7 days after sugery

SECONDARY OUTCOMES:
The incidence of postoperative delirium within 7 days after upper abdominal surgery in patients without liver cirrhosis. | within 7 days after sugery

IPD SHARING:
Plan to Share IPD: Undecided
If the subsequent metabolomics or gut microbiome analyses yield particularly significant findings, these data may initially remain unpublished as they could require further validation through basic animal experiments.